CLINICAL TRIAL: NCT02429999
Title: The Role of Aromatase Inhibitor (Letrozole) in Minimal Ovarian Stimulation Protocols in Assisted Reproductive Technology. A Randomized Controlled Trial
Brief Title: Letrozole in Assisted Reproductive Technology
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, amr shehata abdelbadie, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART
Record Dates: First submitted 2015-04-25; First posted 2015-04-29 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: to Evaluate Letrozole as a Modality for Minimal Ovarian Stimulation in ICSI Cycles .
MeSH Terms: interventions — Ovulation Induction

ARMS (2):
- Letrozole plus FSH (Active Comparator): letrozole, 10 mg daily from day 3-7 and FSH 75 international unit(IU) /day from day 5 continuously and GnRH antagonist (orgalutran 0.25) is given when the follicle size equal to 14 mm till human chorionic gonadotrophin (hCG) injection.
  Interventions: Drug: Letrezole plus FSH
- Standered protocol for induction of ovulation (Active Comparator): 0.1 decapeptyl from day 21 in the previous cycle and continuously stimulated by FSH (150-225 international unit/day) from day 2. We will give them at first 225 international unit FSH for 5 days.
  Interventions: Drug: Standard protocol for induction of ovulation

INTERVENTIONS:
Drug: Letrezole plus FSH — letrozole, 10 mg daily from day 3-7 and FSH 75IU/day from day 5 continuously and GnRH antagonist (orgalutran 0.25) is given when the follicle size equal to 14 mm till hCG injection.
  Arms: Letrozole plus FSH
Drug: Standard protocol for induction of ovulation — 0.1 decapeptyl from day 21 in the previous cycle and continuously stimulated by FSH (150-225IU/day) from day 2.
  Arms: Standered protocol for induction of ovulation

SUMMARY:
Infertility in not a health problem and that infertile couples are not really ill. However, this narrow interpretation of the problem is refuted by the world community. The WHO defines health as a "state of complete physical, mental and social wellbeing and not merely the absence of disease or infirmity". It has also been argued that overpopulation is the main problem in the developing countries and that helping infertile couples contradicts the interests of the countries and the world at large. However, this narrow approach contradicts human rights in general and reproductive rights in particular.

In 1994, the United Nations International Conference on Population and Development in Cairo mentioned issues on future actions on 'prevention and appropriate treatment of infertility where feasible'. However, no guidelines or concrete actions and programmes were given for developing countries.

Worldwide, more than 80 million couples suffer from infertility; the majority of this population are residents of developing countries.

In September 2001, a meeting on 'Medical, Ethical and Social Aspects of Assisted Reproduction' was organized by the WHO. For the first time, major attention was paid to ongoing developments in assisted reproduction technology together with their social and ethical implications in developing countries . It was the first time that the WHO highlighted the issue of assisted reproduction in developing countries.

ART in developed countries is highly expensive one of steps is ovulation induction the most common protocol for induction is the long gonadotrophin-releasing hormone (GnRH) agonist pituitary suppression regimen combined with relatively high doses of exogenous follicle-stimulating hormone (FSH) remains the most frequently used stimulation protocol which is expensive. in our study we will use a mild ovarian stimulating protocol letrozole adjuvant to gonadotrophins which is less expensive

The use of aromatase inhibitor have only recently been introduced in infertility treatment, especially for ovulation induction.

An aromatase inhibitor blocks the conversion of androgens to estrogens in the ovarian follicles, peripheral tissues, and in the brain. This result in two things: (a) Fall in circulating and local estrogens and (b) Rise in intraovarian androgens. Fall in estrogen levels, releases the hypothalamopituitary axis from the negative feedback of estrogens. Thus, there is a surge in follicle stimulating hormone (FSH) release, which results in follicular growth. Since, the feedback mechanism is intact; normal follicular growth, selection of dominant follicle, and atresia of smaller growing follicle occurs; and thereby facilitating monofollicular growth and ovulation.Another mechanism of action of the aromatase inhibitors is by the increasing intraovarian androgens. This increases the follicular sensitivity to FSH. Recent data shows the role of androgens in early follicular developments. by augmenting FSH receptors and stimulating insulin-like growth factor (IGF)-I; FSH and IGF-I act synergistically to promote follicular growth. This pharmacodynamics of letrozole ensures improved endometrial thickness, cervical mucus, monofollicular, and better folliculogenesis. So , these factors may lead to higher pregnancy rates and greater likelihood of singleton pregnancy.

Letrozole has been tried for ovarian stimulation for assisted reproduction. With the concept of mild stimulation in IVF to improve implantation rate, letrozole is a potential agent. Letrozole has two potential uses in IVF: First, where it is used in the follicular phase usually with FSH/human menopausal gonadotropin (HMG) for ovulation induction; second, it has also been used in luteal phase of stimulated IVF cycle and to reduce circulating E2 levels; thus, potentially reducing ovarian hyperstimulation syndrome (OHSS) risk.

A significant reduction in the total dose of gonadotrophins was found when aromatase inhibitor was added in controlled ovarian hyperstimulation (COH) cycles.

Some studies evaluated the addition of letrozole in patients with normal ovarian response undergoing IVF or Intracytoplasmic sperm injection( ICSI). They showed higher implantation and ongoing pregnancy rates in the letrozole cotreatment group.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility.
* Tubal factor. Included treated hydrosalpinx and pyosalpinx
* BMI 18-29.
* Antral follicle count (AFC) more than 5 follicles in one ovary.
* Normal male semen analysis.Mild male factor: concentrations 10 million - 20 million sperm/ml. Moderate male factor : concentrations 5 million - 10 million sperm/ml.

Exclusion Criteria:

* Patients with Endometriosis.
* Azoospermic male.
* BMI more than 29.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
total dose of FSH administered | 2 years
The number of mature follicles developed | 2 years
the levels of terminal E2 pg/mL | 2 years
number of oocytes retrieved | 2 years
endometrial thickness/mm | 2 years
number transferable embryos | 2 years

SECONDARY OUTCOMES:
Number of patient who get pregnant | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- of Medicine, Asyut, Egypt